CLINICAL TRIAL: NCT07167719
Title: Resilience in Reentry: Cognitive-Behavioral Resilience Training for Parolees With Adjustment Challenges
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Massachusetts Institute of Technology (MIT) (Unknown)
Responsible Party: Principal Investigator, Emily Greene Owens, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7520
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Adjustment
Keywords: Incarceration; Reentry
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study employees two arms: the treatment arm and an assessment only arm. The pilot study is non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will receive a 5-session CBT intervention
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Assessment Only (No Intervention): Participants will receive study assessments

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Brief Cognitive-Behavioral Therapy (CBT) focused on building resiliency in response to the effects of institutionalization
  Other Names: CBT
  Arms: Treatment

SUMMARY:
This pilot study assesses the feasibility and acceptability of delivering a brief Cognitive-Behavioral Resiliency treatment to a population of recently released parolees. This study will also give a preliminary indication if the treatment is associated with reliable improvements in adjustment symptoms and well-being for parolees.

DETAILED DESCRIPTION:
In the proposed pilot study, residents of a reentry facility in Los Angeles, CA will be able to enroll in a course of brief (5-session) Cognitive-Behavioral Therapy (CBT) focused on building resiliency in response to the effects of institutionalization. Those who choose to receive the intervention will be included in the intervention group (target N = 30). Those who choose not to receive the intervention will be given the opportunity to complete assessments at the same intervals as the intervention group (assessment only group; target N = 30). Participants will report their degree of satisfaction with the program and how much they think they benefitted from the program at postintervention. Participants will complete self-report measures of adjustment disorder symptoms, flourishing, meaning and purpose in life, and PTSD symptoms at pretreatment (baseline), posttreatment (5 weeks after baseline), and 2-month follow-up (13 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Speaks English
* Been on parole for two years or less.
* Score of 8.5 or higher (range 4 to 16) on the Adjustment Disorder New Module 4 (ADNM-4) screening tool (Ben-Ezra, et al., 2018).

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adjustment Disorder New Module 20 | From pretreatment (baseline) to the end of treatment (5 weeks after baseline)
  The ADNM-20 is a self-report measure consisting of two parts: a stressor list and an item list. It is a 20-item measure that ranges from 20 to 80. Participants will fill out stressors from their prison term and will then complete the items which are composed of a 4-point Likert scales from "Never" to "Often."
Flourishing Scale | From pretreatment (baseline) to the end of treatment (5 weeks after baseline)
  The Flourishing Scale is an 8-item self-report measure (with a range of 8 to 56) of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism. The scale provides a single psychological well-being score.
PROMIS Meaning and Purpose Short Form 8a | From pretreatment (baseline) to the end of treatment (5 weeks after baseline)
  The PROMIS Meaning and Purpose is an 8-item self-report measure with a range of 8 to 40 that assess one's sense of life having purpose and that there are good reasons for living. Higher scores indicate hopefulness, optimism, goal-directedness, and feelings that one's life is worthy.

SECONDARY OUTCOMES:
PTSD Checklist 5 | From pretreatment (baseline) to the end of treatment (5 weeks after baseline)
  This is an 8-item abbreviated version of the PTSD Checklist 5, a self-report measure which ranges from 0 to 32 that assesses the DSM-5 symptoms of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Owens, Study Director — University of California, Irvine
Locations (1):
- The Francisco Homes, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is a small sample size and the study participant's are a systemically vulnerable population.